CLINICAL TRIAL: NCT00248482
Title: Phase II Trial of Imatinib Mesylate Maintenance Therapy in Patients With C-Kit (+) Extensive-Stage Small Cell Lung Cancer
Brief Title: Imatinib Mesylate After Irinotecan and Cisplatin in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000445222; P30CA022453 (NIH); WSU-C-2461 (Other: Barbara Ann Karmanos Cancer Institute); WSU-UMCC-2001-066; CST1571B US93 (Other: Novartis Pharmaceuticals)
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Cisplatin; Imatinib Mesylate; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Irinotecan, Cisplatin & Gleevec™ (Experimental): Cisplatin 60mg/m2 IV day 1 every 21 days x 4 cycles
  Gleevec™ 400 mg po BID (800mg/day)- for patients with objective response or stable disease.
  Irinotecan 65 mg/m2 IV days 1, 8 every 21 days x 4 cycles
  Interventions: Drug: Cisplatin; Drug: Gleevec™; Drug: irinotecan

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 60mg/m2 IV day 1 every 21 days x 4 cycles
  Other Names: Platinol ®; Platinol®-AQ; CDDP
Drug: Gleevec™ — Gleevac 400 mg po BID (800mg/day)- fo patients with objective response or stable disease.
  Other Names: STI-571; imatinib mesylate
Drug: irinotecan — Irinotecan: 65 mg/m2 IV days 1, 8 every 21 days x 4 cycles
  Other Names: Camptosar®; Camptothecin-11; CPT-11

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as irinotecan and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Giving imatinib mesylate after irinotecan and cisplatin may keep the tumor from coming back.

PURPOSE: This phase II trial is studying how well giving imatinib mesylate after irinotecan and cisplatin works in treating patients with extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 4-month progression-free survival rate in patients with c-kit positive, extensive stage small cell lung cancer treated with maintenance therapy comprising imatinib mesylate after induction therapy comprising irinotecan and cisplatin.

Secondary

* Determine the overall survival of patients treated with this regimen.
* Determine the tolerability of imatinib mesylate maintenance therapy in these patients.
* Determine the response rate in patients treated with irinotecan and cisplatin.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive irinotecan IV over 90 minutes on days 1 and 8 and cisplatin IV on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a response (partial or complete) or stable disease proceed to maintenance therapy.
* Maintenance therapy: Patients receive oral imatinib mesylate twice daily for 6 months in the absence of disease progression or unacceptable toxicity. Some patients may continue to receive therapy for up to 1 year.

After completion of study treatment, patients are followed for 4 months.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell lung cancer (SCLC)

  * Extensive stage disease, defined by 1 of the following criteria:

    * Disease extends beyond one hemithorax and regional lymph nodes
    * Cytologically positive pleural effusion
* Meets 1 of the following criteria:

  * Measurable disease, defined as ≥ 1 unidimensionally measurable lesion outside the field of any prior radiotherapy
  * Evaluable disease
* No history of untreated or symptomatic brain or leptomeningeal metastases

  * Prior brain metastases allowed provided patient is neurologically stable for 2 weeks after completion of therapy

PATIENT CHARACTERISTICS:

Performance status

* SWOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8 g/dL

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Meets 1 of the following criteria:

  * Alkaline phosphatase (AP) normal AND AST and ALT ≤ 2.5 times ULN
  * AP ≤ 5 times ULN AND AST and ALT normal
* No acute or chronic liver disease (e.g., chronic active hepatitis or cirrhosis)

Renal

* Creatinine normal OR
* Creatinine clearance ≥ 65 mL/min

Cardiovascular

* No uncontrolled congestive heart failure
* No uncontrolled angina
* No myocardial infarction and/or stroke within the past 3 months

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No peripheral neuropathy ≥ grade 2
* No symptomatic edema from any etiology
* No known HIV positivity
* No other serious medical illness
* No other malignancy within the past 3 years except adequately treated squamous cell or basal cell skin cancer or carcinoma in situ of the cervix
* No history of dementia, active psychiatric disorder, or other condition that would preclude study compliance or ability to take oral medication on a daily basis

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No prior chemotherapy for SCLC

Endocrine therapy

* No concurrent routine systemic corticosteroids

Radiotherapy

* See Disease Characteristics
* At least 2 weeks since prior palliative radiotherapy

Surgery

* More than 2 weeks since prior major surgery

Other

* No concurrent therapeutic anticoagulation with warfarin

  * Concurrent low molecular weight heparin allowed provided regimen was initiated ≥ 2 weeks prior to study entry
* No other concurrent participation in another study of an investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2002-02; Primary Completion 2005-04 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | at 4 months

SECONDARY OUTCOMES:
Overall survival | at least 4 months after discontinuation of treatment
Tolerability of Gleevec maintenance therapy | 30 days after completion of study treatment
Response rate as measured by RECIST at | Baseline and every 8 weeks during study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shirish M. Gadgeel, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (2):
- United States (2):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan